CLINICAL TRIAL: NCT05779189
Title: Effects of Game-based Virtual Reality Intervention on Senior Fitness, Fall Prevention and Balance Function Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202204048
Record Dates: First submitted 2023-03-03; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-05

CONDITIONS: Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive conventional health education and game-based virtual reality (game) in person.
  Interventions: Behavioral: Game-based virtual reality (Game)
- Control (Active Comparator): Participants will receive conventional health education and 4 video of balance exercise.
  Interventions: Behavioral: Conventional health education

INTERVENTIONS:
Behavioral: Game-based virtual reality (Game) — Besides reading the health education flier, they also need to trained with the game-based virtual reality in Biodex Medical Systems, which is a machine, includes 4 games: Catch Game, boating, Ball Maze, and Word Search. And all of the games are balance control games. The games were implemented in person for 30 minutes one time, total is 16 times (once to twice day a week).
  Arms: Intervention
Behavioral: Conventional health education — The health education flier was made refer to medical institutions, e.g., hospitals or clinics, the video of balance exercise was collected from the internet. Participants were assigned to read the health education flier, and follow suit the video of balance exercise at home of their free will.
  Arms: Control

SUMMARY:
The purpose of this study is to explore the effectiveness between game-based virtual reality intervention and conventional health education in improving older adults' balance knowledge, and let them know how to prevent falling. The intervention group will receive virtual reality games in person and read the health education flier, while the control group was assigned to read the health education flier and follow suit the video of balance exercise.

DETAILED DESCRIPTION:
Falls can lead to disability, sickbed and even death of the elderly, and it ranks second among the top ten which causes death in Taiwan. In the past, when multifaceted exercise interventions were conducted for the elderly, most of them focused on group strength training and aerobic exercise, but lacked individualized balance training, resulting in a low degree of cooperation.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people over the age of 65-99.

Exclusion Criteria:

* cognitive impairment
* neurological diseases
* severe osteoporosis
* lower limb joint surgery
* discomfort symptoms during exercise

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test | Right after the intervention
  Participants were assigned to do 2 tasks of the test. One is time up and go, and the other one is eyes-open single-leg stance test. We recorded the time (in seconds) they took.
Falls Efficacy Scale International | Right after the intervention
  Participants were assessed by the questionnaire, and we recorded the points of the participants. The higher the point is, the more concerned they are about the falls.
Balance or sensory-Integration test | Right after the intervention
  The balance of postural-stability test and the modified clinical test of sensory integration and balance (m-CTSIB) were performed using the Biodex Stability System (BSS; Biodex Medical Systems, Shirley, New York, USA).
Balance of postural-stability test | Right after the intervention
  The balance of postural stability was tested according to 3 stability indices (overall stability; anterior-to-posterior stability; and medial-to-lateral stability).
Modified Clinical Test for Sensory Integration of Balance (m-CTSIB) | Right after the intervention
  The m-CTSIB, which includes 4 sway indices, was conducted 4 sensory conditions: (1) eyes open whilst standing on a firm surface (EOFIS); (2) eyes closed whilst standing on a firm surface (ECFIS): (3) eves open whilst standing on an unstable (foam) surface (EOFOS); and (4) eyes closed whilst standing on an unstable (foam) surface (ECFOS).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei County, Taiwan